CLINICAL TRIAL: NCT02305927
Title: Trial of Vitamin D in HIV Progression, Birth Outcomes, and Child Health
Acronym: ToV5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wafaie Fawzi (Other)
Collaborators: Management and Development for Health (MDH) (Unknown)
Responsible Party: Sponsor-Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Organization: Harvard School of Public Health (HSPH) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01HD083113 (NIH)
Record Dates: First submitted 2014-10-29; First posted 2014-12-03 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: HIV
Keywords: Vitamin D; Pregnant women
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (cholecalciferol) (Experimental)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — Supplements containing 3,000 IU vitamin D3 taken orally once per day by the mother starting from the second trimester until 12 months postpartum
  Arms: Vitamin D3 (cholecalciferol)
Other: Placebo — Placebo supplements taken orally once per day by the mother starting from the second trimester until 12 months postpartum
  Arms: Placebo

SUMMARY:
The purpose of this study to assess the effect of maternal vitamin D3 (cholecalciferol) supplementation on maternal HIV progression, small-for-gestational age infants, and infant stunting at 12 months postpartum for HIV-infected Tanzanian pregnant women who are receiving highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled trial of maternal vitamin D3 (cholecalciferol) supplementation starting in the second trimester (12-27 weeks gestation) and continuing until 12 months postpartum among HIV-infected Tanzanian pregnant women who are receiving HAART. Eligible individuals are randomized to receive a) a vitamin D3 regimen consisting 3,000 IU of vitamin D3 taken orally once daily starting in the second trimester and continuing until 12 months postpartum or b) a placebo regimen taken orally once daily starting in the second trimester and continuing until 12 months postpartum. Mothers will be followed at study visits during pregnancy and mother/infant pairs will attend study visits from birth until trial discharge at 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years old
* HIV-positive
* Receiving HAART
* Pregnant and of 12-27 weeks gestation (Second Trimester)
* Calcium levels in the normal physiologic range (≤2.6 mmol/L)

Exclusion Criteria:

* Enrolled in any other clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Proportion of participants experiencing maternal HIV progression | Second Trimester until 12 months post partum
Proportion of small-for-gestational age infants | Birth
Proportion of stunted infants (height-for-age z-score < -2) | 12 months postpartum (1 year of age)

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Christopher R Sudfeld, ScD, Principal Investigator — Harvard School of Public Health (HSPH); Karim P Manji, MD, Principal Investigator — Management and Development for Health (MDH)
Locations (1):
- Management and Development for Health (MDH), Dar es Salaam, Tanzania

REFERENCES:
- [Background] Sudfeld CR, Manji KP, Duggan CP, Aboud S, Muhihi A, Sando DM, Al-Beity FMA, Wang M, Fawzi WW. Effect of maternal vitamin D3 supplementation on maternal health, birth outcomes, and infant growth among HIV-infected Tanzanian pregnant women: study protocol for a randomized controlled trial. Trials. 2017 Sep 4;18(1):411. doi: 10.1186/s13063-017-2157-3. PMID 28870263
- [Derived] Shobanke T, Muhihi A, Perumal N, Ulenga N, Al-Beity FMA, Duggan CP, Fawzi WW, Manji KP, Sudfeld CR. Effect of vitamin D supplementation during pregnancy and lactation on the development of infants born to Tanzanian women living with HIV: a secondary analysis of a randomised controlled trial. BMJ Open. 2025 Oct 20;15(10):e098723. doi: 10.1136/bmjopen-2024-098723. PMID 41120170
- [Derived] Lauer JM, Kirby MA, Muhihi A, Ulenga N, Aboud S, Liu E, Choy RK, Arndt MB, Kou J, Fawzi WW, Gewirtz AT, Sudfeld CR, Manji KP, Duggan CP. Effects of Vitamin D-3 Supplementation During Pregnancy and Lactation on Maternal and Infant Biomarkers of Environmental Enteric Dysfunction, Systemic Inflammation, and Growth: A Secondary Analysis of a Randomized Controlled Trial. J Nutr. 2024 Nov;154(11):3400-3406. doi: 10.1016/j.tjnut.2024.08.032. Epub 2024 Sep 13. PMID 39278411
- [Derived] Sudfeld CR, Manji KP, Muhihi A, Duggan CP, Aboud S, Alwy Al-Beity FM, Wang M, Zhang N, Ulenga N, Fawzi WW. Vitamin D3 supplementation during pregnancy and lactation for women living with HIV in Tanzania: A randomized controlled trial. PLoS Med. 2022 Apr 15;19(4):e1003973. doi: 10.1371/journal.pmed.1003973. eCollection 2022 Apr. PMID 35427363